CLINICAL TRIAL: NCT02617992
Title: Systematic Wide-Field EMR Scar Assessment and Therapy Audit
Acronym: SANT
Status: Completed | Type: Observational
Sponsor: Western Sydney Local Health District (Other)
Responsible Party: Principal Investigator, Professor Michael Bourke, Director of Gastrointestinal Endoscopy, Western Sydney Local Health District
Other Study IDs: HREC2013/8/6.5 (3796)
Record Dates: First submitted 2015-11-08; First posted 2015-12-01 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Polyps
MeSH Terms: conditions — Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- EMR Surveillance: Patients who are referred for Endoscopic Mucosal Resection of Upper Gastrointestinal Lesions undertaking a surveillance visit will be included in this cohort.

SUMMARY:
The development of a standardised imaging protocol to detect post endoscopic mucosal resection (EMR) recurrence or residual adenoma through the comparison of biopsies of the post EMR scar with endoscopic findings.

DETAILED DESCRIPTION:
Removal of colonic polyps reduces colon cancer and although most polyps found are small, removal of large polyps can now be safely and effectively removed with wide field EMR. Residual polyp tissue is found at follow up colonoscopy in approximately 15% of cases however and remains a focus of attempts to improve EMR efficacy. All patients undergoing surveillance colonoscopy after EMR at Westmead Hospital Endoscopy unit will have steps of assessment and therapy of the scar recorded. Data will be entered into the large prospective audit database and also analysed separately. Data will be stored in coded format. The individual steps and the outcome of the scar interrogation and therapy will also be assessed and analysed. It is expected that these results will help guide the optimal approach to assessment and confirm the efficacy of therapy of recurrence further aiding the endoscopic approach to large colonic polyps.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surveillance colonoscopy of a previously resected large sessile colonic polyp or laterally spreading tumour ≥20mm in size.
* Age > 18 years
* Able to give informed consent to involvement in the clinical study

Exclusion Criteria:

* Unable to provide informed consent for involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had endoscopic mucosal resection of colonic polyps that are undergoing surveillance colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Presence of post-EMR recurrence | one year
  Presence of post-EMR recurrence

SECONDARY OUTCOMES:
Histological characteristics of post-EMR scar biopsies | one year
Scar size | one year
  Scar size (maximum dimension)
Presence of post EMR scar with clip artifact | one year
  Presence of post EMR scar with clip artifact, recognized as one or more nodule within the scar with a normal pit pattern
Number of sites of recurrence | one year
  Number of sites of recurrence (unifocal, 2 sites, 3 or more sites)
Location of recurrence | one year
  Location of recurrence (edge of the scar, within the scar or both)
Morphology of recurrence | one year
  Morphology of recurrence (flat or elevated)
Kudo pit pattern assessment | one year
  Kudo pit pattern and whether the pit pattern of recurrence is only seen with NBI
NICE classification | one year
  As recurrence is diminutive the NICE classification is also applied and so the NBI appearance of recurrence (darker or lighter than the scar) is noted.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bourke, MBBS, Principal Investigator — Western Sydney Local Health District
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia